CLINICAL TRIAL: NCT01332149
Title: An 11-week Randomized, Double-blind, Multi Center, Placebo-controlled Study To Evaluate The Efficacy, Safety And Tolerability Of Pregabalin (300 Mg/Day) Using A Fixed Dosing Schedule In The Treatment Of Subjects S With Pain Associated With Diabetic Peripheral Neuropathy.
Brief Title: Study To Evaluate Efficacy, Safety And Tolerability Of Lyrica In Patients With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081265
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-06

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetic Neuropathies; Pain; Efficacy of pregabalin; Placebo controlled
MeSH Terms: conditions — Diabetic Neuropathies; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 300 mg/day pregabalin (Lyrica) (Experimental): Patient take pregabalin capsule twice a day
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matched with pregabalin

INTERVENTIONS:
Drug: Pregabalin — Subjects in the pregabalin group will start treatment with pregabalin capsule 150 mg/day for 1 week, then their dose will be increased to 300mg/day. After 1-week titration period, dose must be stable during study, no dose adjustment is permitted, and subject who cannot tolerate 300 mg/day pregabalin will be withdrawn.
  At the completion of the dose maintenance phase subjects will taper off study medication over a 1-week period. 300 mg/ day subjects will taper to 150 mg/ day.
  Arms: 300 mg/day pregabalin (Lyrica)
Drug: Placebo matched with pregabalin — Subject will take placebo matched with pregabalin twice a day.
  Arms: Placebo

SUMMARY:
Pregabalin has proven effective in previous clinical trails in other countries in relieving neuropathic pain associated with postherpetic neuralgia and painful diabetic neuropathy.

This study is being conducted according to China registration requirement to submit a reapplication with new local diabetic peripheral neuropathy study as a commitment plus the existing data to apply for Lyrica "pain associated with postherpetic neuralgia" indication after Lyrica "pain associated with postherpetic neuralgia" is approved.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years or older
* Diagnosis of painful, distal, symmetrical, sensorimotor polyneuropathy which is due to diabetes mellitus (Type 1 or 2), and symptoms of painful diabetic neuropathy for 6 months to 5 years (inclusive).
* At the baseline and randomization visits, a score of ≥50 mm on the Visual Analogue Scale, at randomization, subjects must have completed at least 5 daily pain interference diaries, and have an average daily pain score of ≥5 over the past 7 days.
* Patient who are willing and capable to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Women of childbearing potential are willing to use contraception during study.

Exclusion Criteria:

* Subjects with more than 30% decrease on the Pain Visual Analog Scale at randomization as compared to screening; and during the 1 week screening period, with more than one pain score <3 in pain scores.
* Subject has other kinds of neurological disorder, pain of other reason, or skin condition that could confuse the assessment.
* Subject with any other serious or unstable condition which in the opinion of the investigator might compromise participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- China (30):
  - Southwest hospital of the third military medical university/Department of Neurology, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - Department of Endocrinology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Dept. of Endocrinology, The first Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Dept. of Endocrinology, The second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital,Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - Xiangya Hospital of Centre-south University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Dept. of Endocrinology, The second hospital of Jilin University, Changchun, Jilin
  - Shengjing hospital of china medical university, Shenyang, Liaoning
  - Qilu Hospital of Shandong University/department of internal neurology, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of medicine, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Tiantan Hospital affiliated to Capital Medical University, Neurology Department, Beijing
  - Peking University Third Hospital, Beijing
  - Endocrinology Department, Beijing
  - Beijing Hospital of the Ministry of Health, Beijing
  - Tongren Hospital Affiliated to Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - GuangZhou First Municipal People's Hospital, Guangzhou
  - Shanghai Changzheng Hospital, Shanghai
  - Huashan Hospital Affiliated Fudan University, Neurology Department, Shanghai
  - Shanghai Tenth People's Hospital/The Endocrinology Department, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Renji Hospital Shanghai Jiao Tong University School of Medicine/Neurology Department, Shanghai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081265&StudyName=Study%20To%20Evaluate%20Efficacy%2C%20Safety%20And%20Tolerability%20Of%20Lyrica%20In%20Patients%20With%20Painful%20Diabetic%20Peripheral%20Neuropathy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were Chinese. 626 participants were randomized initially, as originally stated on clinicaltrials.gov. However, 3 participants discontinued right after randomization without any treatment information. As such, the actual number of participants randomized and assigned to treatment was 623 as stated in the "Started" Row below.
Groups:
- Pregabalin: Participants received 1 placebo capsule matched to pregabalin twice a day for 1 week (run-in period), followed by a 9-week double-blind treatment phase (1-week dose-escalation phase where participants received pregabalin 150 milligram [mg] per day in the form of 75 mg twice a day and an 8-week fixed dose phase where participants received pregabalin 300 mg per day in the form of 150 mg twice a day), and a 1-week taper-off phase where participants received pregabalin 150 mg per day (in the form of 75 mg twice a day).
- Placebo: Participants received matching placebo capsule(s) for a period of 11 weeks， which consisted of a 1-week run-in period, 9-week double-blind treatment phase and 1-week taper-off period.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 314 (Assigned to study treatment.) | 309 (Assigned to study treatment.)
Treated | 313 | 307
Completed | 284 | 271
Not Completed | 30 | 38
Not completed — Adverse Event | 11 | 9
Not completed — Other unspecified | 5 | 7
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Insufficient clinical response | 4 | 7
Not completed — Did not meet entrance criteria | 3 | 4
Not completed — Randomized but not treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 313 | 307 | 620
Age, Customized [Number; unit: participants]
  18-44 years | 25 (10.3) | 15 (9.5) | 40
  45-64 years | 172 | 178 | 350
  More than or equal to (>=) 65 years | 116 | 114 | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 168 | 327
  Male | 154 | 139 | 293

OUTCOME MEASURES:

1. Primary Outcome: Baseline Mean Pain Score
Description: The daily pain rating scale (DPRS) consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10.
Time Frame: Baseline
Population: All participants in the Full Analysis Set (FAS) population, consisting of all participants randomized to treatment that received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale | 6.65 (1.117) | 6.67 (1.150)

2. Primary Outcome: Change From Baseline in Mean Pain Score at Endpoint
Description: The daily pain rating scale (DPRS) consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. The mean endpoint pain score was obtained from the last 7 available DPRS scores of the daily pain diary while the participant was on study medication, up to and including the day after the last Week 8 (Day 57) dose.
Time Frame: Baseline and end of fixed dose phase (Day 63/Week 9)/Early Termination (Study Endpoint)
Population: All participants in the Full Analysis Set (FAS) population (all participants randomized to treatment that received at least 1 dose of study medication) who had available data for this outcome measure. The Last Observation Carried Forward (LOCF) method was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 312 | 307
units on a scale | -2.14 (0.115) | -1.86 (0.117)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0559, ANCOVA — Primary analysis was two-sided and performed at the 0.05 significance level. No multiple comparisons adjustment was made; The ANCOVA model included treatment and study center as factors and the corresponding baseline score as a covariate in the model; Least Squares (LS) Mean Difference = -0.28, 95% CI 2-sided [-0.58 to 0.01], Standard Error of Mean 0.148

3. Secondary Outcome: Change From Baseline in Weekly Mean Pain Score at Weeks 1 to 9
Description: The DPRS consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. The weekly mean pain score was the sum of the daily scores divided by the number of diary entries during that week. The overall change is the average change from Weeks 1 to 9.
Time Frame: Baseline and weekly from Weeks 1 to 9
Population: The FAS population consisted of all participants randomized to treatment that received at least 1 dose of study medication. N=number of evaluable participants at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale
  Week 1 change from baseline (N=312, 307) | -0.60 (0.091) | -0.36 (0.092)
  Week 2 change from baseline (N=304, 295) | -0.97 (0.092) | -0.71 (0.093)
  Week 3 change from baseline (N=298, 291) | -1.25 (0.092) | -1.01 (0.093)
  Week 4 change from baseline (N=297, 289) | -1.47 (0.092) | -1.21 (0.093)
  Week 5 change from baseline (N=296, 287) | -1.61 (0.092) | -1.39 (0.093)
  Week 6 change from baseline (N=293, 278) | -1.84 (0.092) | -1.59 (0.094)
  Week 7 change from baseline (N=290, 275) | -2.04 (0.092) | -1.77 (0.094)
  Week 8 change from baseline (N=290, 275) | -2.18 (0.092) | -1.88 (0.094)
  Week 9 change from baseline (N=287, 273) | -2.32 (0.092) | -2.07 (0.094)
  Overall change from baseline | -1.59 (0.082) | -1.33 (0.083)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0527, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.23, 95% CI 2-sided [-0.47 to 0.00], Standard Error of Mean 0.120
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0279, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.27, 95% CI 2-sided [-0.50 to -0.03], Standard Error of Mean 0.121
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0508, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.24, 95% CI 2-sided [-0.48 to 0.00], Standard Error of Mean 0.121
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0349, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.26, 95% CI 2-sided [-0.49 to -0.02], Standard Error of Mean 0.121
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0672, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.22, 95% CI 2-sided [-0.46 to 0.02], Standard Error of Mean 0.122
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0469, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.24, 95% CI 2-sided [-0.48 to -0.00], Standard Error of Mean 0.122
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 7 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0280, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.27, 95% CI 2-sided [-0.51 to -0.03], Standard Error of Mean 0.122
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0140, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.30, 95% CI 2-sided [-0.54 to -0.06], Standard Error of Mean 0.122
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Week 9 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0375, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.25, 95% CI 2-sided [-0.49 to -0.01], Standard Error of Mean 0.122
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Overall change from baseline analysis. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0164, Mixed Model Repeated Measures Analysis — All analyses were two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.25, 95% CI 2-sided [-0.46 to -0.05], Standard Error of Mean 0.105 — Overall change was estimated from the mixed effect model treatment main effect

4. Secondary Outcome: Baseline Mean Sleep Interference Score
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale | 5.25 (2.236) | 5.12 (2.278)

5. Secondary Outcome: Change From Baseline in Mean Sleep Interference Score at Endpoint
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10. The mean endpoint score was obtained from the last 7 available scores of the daily diary while the participant was on study medication, up to and including the day after the last Week 9 (Day 63) dose.
Time Frame: Baseline and end of fixed dose phase (Day 63/Week 9)/Early Termination (Study Endpoint)
Population: All participants in the FAS population (all participants randomized to treatment that received at least 1 dose of study medication) who had available data for this outcome measure. The LOCF method was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 311 | 307
units on a scale | -1.52 (0.110) | -1.30 (0.112)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1340, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.21, 95% CI 2-sided [-0.49 to 0.07], Standard Error of Mean 0.143

6. Secondary Outcome: Change From Baseline in Weekly Mean Sleep Interference Score at Weeks 1 to 9
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10. The weekly mean score was the sum of the daily scores divided by the number of diary entries during that week. The overall change is the average change from Weeks 1 to 9.
Time Frame: Baseline and weekly from Weeks 1 to 9
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale
  Week 1 change from baseline (N=311, 307) | -0.38 (0.096) | -0.26 (0.098)
  Week 2 change from baseline (N=303, 295) | -0.66 (0.097) | -0.51 (0.098)
  Week 3 change from baseline (N=297, 291) | -0.88 (0.097) | -0.72 (0.099)
  Week 4 change from baseline (N=296, 289) | -1.06 (0.097) | -0.86 (0.099)
  Week 5 change from baseline (N=295, 287) | -1.14 (0.097) | -0.98 (0.099)
  Week 6 change from baseline (N=292, 278) | -1.32 (0.098) | -1.07 (0.099)
  Week 7 change from baseline (N=289, 275) | -1.43 (0.098) | -1.25 (0.099)
  Week 8 change from baseline (N=289, 275) | -1.59 (0.098) | -1.36 (0.099)
  Week 9 change from baseline (N=286, 273) | -1.67 (0.098) | -1.49 (0.100)
  Overall change from baseline | -1.13 (0.085) | -0.94 (0.087)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3438, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.12, 95% CI 2-sided [-0.37 to 0.13], Standard Error of Mean 0.127
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.2482, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.15, 95% CI 2-sided [-0.40 to 0.10], Standard Error of Mean 0.128
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.2249, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.16, 95% CI 2-sided [-0.41 to 0.10], Standard Error of Mean 0.129
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.1094, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.21, 95% CI 2-sided [-0.46 to 0.05], Standard Error of Mean 0.129
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.2095, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.16, 95% CI 2-sided [-0.41 to 0.09], Standard Error of Mean 0.129
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 6]; Test type: Superiority or Other; p = 0.0531, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.25, 95% CI 2-sided [-0.50 to 0.00], Standard Error of Mean 0.129
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.1628, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.18, 95% CI 2-sided [-0.44 to 0.07], Standard Error of Mean 0.130
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 8]; Test type: Superiority or Other; p = 0.0770, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.23, 95% CI 2-sided [-0.48 to 0.02], Standard Error of Mean 0.130
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.1651, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.18, 95% CI 2-sided [-0.43 to 0.07], Standard Error of Mean 0.130
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 10]; Test type: Superiority or Other; p = 0.1006, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.18, 95% CI 2-sided [-0.40 to 0.04], Standard Error of Mean 0.110

7. Secondary Outcome: Percentage of 30 Percent (%) Responders at Endpoint
Description: The DPRS consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. A 30% responder was a participant who had 30% reduction or more in mean pain score at the end of the fixed dose phase (Day 63/Week 9) (Study Endpoint) compared to baseline.
Time Frame: End of fixed dose phase (Day 63/Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 312 | 307
percentage of participants | 50.3 (0.115) | 44.3 (0.117)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1309, Cochran-Mantel-Haenszel — Analysis was two-sided and performed at the 0.05 significance level; Cochran-Mantel-Haenszel test comparing pregabalin to placebo adjusted for center; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.93 to 1.74]

8. Secondary Outcome: Change From Baseline in Short Form McGill Pain Questionnaire (SF-MPQ) Score at Weeks 1, 5, and 9
Description: SF-MPQ was assessed according to the participant's answer to the SF-MPQ questionnaire. The score for each composite scale (sensory, affective, and total) was derived by summing the reported intensity value for each item within a particular scale where None=0, Mild=1, Moderate=2, and Severe=3. The sensory score was the sum of the scores of the first 11 pain descriptors (throbbing, shooting, stabbing, sharp, cramping, gnawing, hot-burning, aching, heavy, tender, and splitting) and could range from 0-33. The affective score was the sum of the scores of the last 4 pain descriptors (tiring-exhausting, sickening, fearful, and punishing-cruel) and could range from 0-12. The total score was the sum of the scores of all 15 pain descriptors and could range from 0 to 45. Higher scores indicated greater pain.
Time Frame: Baseline; Weeks 1, 5, and 9
Population: The FAS population consisted of all participants randomized to treatment that received at least 1 dose of study medication. N=number of evaluable participants at the specified time point. No inferential analyses were performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale
  Sensory score, Baseline (N=313, 306) | 7.90 (5.101) | 8.11 (5.098)
  Sensory score, Week 1 change (N=311, 304) | -1.50 (3.422) | -1.34 (3.134)
  Sensory score, Week 5 change (N=297, 288) | -2.89 (4.244) | -2.47 (3.925)
  Sensory score, Week 9 change (N=288, 274) | -3.87 (4.432) | -3.37 (4.348)
  Affective score, Baseline (N=313, 307) | 1.25 (1.809) | 1.20 (1.817)
  Affective score, Week 1 change (N=311, 304) | -0.41 (1.569) | -0.37 (1.410)
  Affective score, Week 5 change (N=297, 289) | -0.72 (1.724) | -0.62 (1.652)
  Affective score, Week 9 change (N=287, 274) | -0.75 (1.744) | -0.62 (1.792)
  Total score, Baseline (N=313, 307) | 9.15 (6.118) | 9.28 (6.445)
  Total score, Week 1 change (N=311, 305) | -1.92 (4.260) | -1.70 (3.908)
  Total score, Week 5 change (N=297, 289) | -3.61 (5.084) | -3.07 (4.893)
  Total score, Week 9 change (N=288, 274) | -4.62 (5.272) | -4.00 (5.512)

9. Secondary Outcome: Baseline Pain Visual Analogue Scale (VAS) and Present Pain Intensity (PPI) Scale
Description: The VAS was part of the Short Form McGill Pain Questionnaire (SF-MPQ) scale and reflected the overall pain intensity score, The pain VAS was a horizontal line; 100 millimeters (mm) in length, was self-administered by the participant in order to rate pain from 0 (no pain) to 100 (worst possible pain). The PPI was part of the SF-MPQ scale and measured the participant's present pain intensity on a 6-point scale ranging from 0 (no pain) to 5 (excruciating).
Time Frame: Baseline
Population: All participants in the FAS population, consisting of all participants randomized to treatment that received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale
  VAS | 69.08 (11.474) | 69.06 (11.811)
  PPI | 2.28 (0.784) | 2.27 (0.830)

10. Secondary Outcome: Change From Baseline in Pain VAS From the SF-MPQ at Endpoint
Description: The VAS was part of the SF-MPQ scale and reflected the overall pain intensity score. The pain VAS was a horizontal line; 100 mm in length, was self-administered by the participant in order to rate pain from 0 (no pain) to 100 (worst possible pain).
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 310 | 304
units on a scale | -25.07 (1.260) | -21.82 (1.279)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0463, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -3.25, 95% CI 2-sided [-6.45 to -0.05], Standard Error of Mean 1.628

11. Secondary Outcome: Change From Baseline in PPI Scale From the SF-MPQ at Endpoint
Description: The PPI was part of the SF-MPQ scale and measured the participant's present pain intensity on a 6-point scale ranging from 0 (no pain) to 5 (excruciating).
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 309 | 305
units on a scale | -0.80 (0.047) | -0.73 (0.048)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.2748, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.07, 95% CI 2-sided [-0.19 to 0.05], Standard Error of Mean 0.061

12. Secondary Outcome: Baseline Medical Outcomes Study (MOS)-Sleep Scale Scores
Description: The MOS-Sleep Scale was a participant-rated instrument which assesses sleep quantity and quality with 12 items (7 subscale scores: sleep disturbance, snoring, awakening short of breath/with headache, sleep adequacy, somnolence, sleep quantity, optimal sleep; and a 9-item overall sleep problems index). Subscale scores total range: 0-100 (except sleep quantity [range 0-24 hours], optimal sleep [yes:1, no:0]). Higher scores=poorer sleep outcomes (except sleep quantity, adequacy, and optimal sleep).
Time Frame: Baseline
Population: All participants in the FAS population (all participants randomized to treatment that received at least 1 dose of study medication) who had available data for this outcome measure. N=number of evaluable participants for each category
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale
  Sleep disturbance score (N=313, 307) | 36.29 (24.768) | 35.13 (26.915)
  Snoring score (N=312, 307) | 35.13 (36.670) | 37.59 (37.163)
  Awaken short of breath score (N=313, 307) | 11.50 (21.557) | 10.75 (21.883)
  Quantity of sleep score (N=311, 304) | 6.07 (2.882) | 5.98 (1.451)
  Sleep adequacy score (N=313, 307) | 57.32 (31.518) | 60.88 (30.274)
  Somnolence score (N=312, 307) | 33.87 (20.459) | 36.03 (21.491)
  Sleep problems index score (N=312, 307) | 32.19 (19.806) | 31.21 (20.388)

13. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Sleep Disturbance Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. For sleep disturbance, the subscale score also ranged from 0 to 100, with higher scores representing greater sleep disturbance.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 297 | 286
units on a scale | -9.11 (1.222) | -7.98 (1.244)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4758, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.13, 95% CI 2-sided [-4.22 to 1.97], Standard Error of Mean 1.577

14. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Snoring Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The snoring subscale score also ranged from 0 to 100, with lower scores indicating less snoring.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 295 | 285
units on a scale | 2.78 (1.716) | -0.53 (1.743)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1363, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 3.31, 95% CI 2-sided [-1.05 to 7.67], Standard Error of Mean 2.220

15. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Awaken Short of Breath Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The awaken short of breath subscale also ranged from 0 to 100, with lower scores indicating less difficulty in breathing.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 295 | 286
units on a scale | -2.10 (1.061) | -2.31 (1.078)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.8808, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.21, 95% CI 2-sided [-2.49 to 2.90], Standard Error of Mean 1.371

16. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Quantity of Sleep Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The MOS Sleep Quantity sub-scale scores ranged from 0 to 24 (number of hours slept).
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 295 | 280
units on a scale | 0.33 (0.085) | 0.14 (0.087)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0887, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.19, 95% CI 2-sided [-0.03 to 0.40], Standard Error of Mean 0.110

17. Secondary Outcome: Percentage of Participants Who Had Optimal Sleep at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The MOS optimal sleep subscale was a binary outcome derived from the sleep quantity responses: the response was YES if sleep quantity was 7 or 8 hours per night.
Time Frame: Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 297 | 282
percentage of participants | 43.8 (0.085) | 45.0 (0.087)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a logistic regression model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.7929, Regression, Logistic — Analysis was two-sided and performed at the 0.05 significance level; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.72 to 1.53]

18. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Sleep Adequacy Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The sleep adequacy subscale also ranged from 0 to 100, with higher scores indicating greater sleep adequacy.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 297 | 285
units on a scale | 8.87 (1.532) | 7.82 (1.552)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.5960, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.05, 95% CI 2-sided [-2.83 to 4.92], Standard Error of Mean 1.973

19. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Somnolence Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The somnolence subscale score also ranged from 0 to 100, with lower scores indicating less somnolence.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 295 | 285
units on a scale | -1.22 (1.187) | -0.88 (1.208)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.8216, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.35, 95% CI 2-sided [-3.36 to 2.67], Standard Error of Mean 1.536

20. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Sleep Problems Index Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The sleep problems index subscale score also ranged from 0 to 100, with lower scores indicating fewer sleep problems.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 294 | 284
units on a scale | -6.71 (0.914) | -5.88 (0.927)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4829, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.83, 95% CI 2-sided [-3.14 to 1.49], Standard Error of Mean 1.177

21. Secondary Outcome: Clinical Global Impression of Change (CGIC) at Endpoint
Description: The CGIC was a clinician-rated global measure that provided a clinically relevant and easy to interpret account of a clinician's perception of the clinical importance of the participant's improvement or worsening during their involvement in a clinical study. Clinicians rated the participant's overall improvement on a 7-point scale where scores ranged from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 299 | 290
units on a scale | 2.58 (0.057) | 2.73 (0.058)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors; Test type: Superiority or Other; p = 0.0431, ANOVA — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.15, 95% CI 2-sided [-0.29 to -0.00], Standard Error of Mean 0.073

22. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Endpoint
Description: The PGIC was a participant-rated global measure that provided a clinically relevant and easy to interpret account of a participant's perception of the clinical importance of their own improvement or worsening during their involvement in a clinical study. Participants rated their overall improvement on a 7-point scale where scores ranged from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 297 | 290
units on a scale | 2.60 (0.057) | 2.74 (0.058)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors; Test type: Superiority or Other; p = 0.0602, ANOVA — Analysis was two-sided and performed at the 0.05 significance level; LS Mean Difference = -0.14, 95% CI 2-sided [-0.28 to 0.01], Standard Error of Mean 0.074

23. Secondary Outcome: Baseline Hospital Anxiety and Depression Scale (HADS) Scores
Description: The HADS was a self-administered questionnaire that consisted of 2 subscales, 1 measuring anxiety (HADS-A Scale) and the other measuring depression (HADS-D Scale). Each subscale comprised of 7 items; participants assessed how each item applied to them on a scale of 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Subscores from HADS-A (Anxiety) and HADS-D (Depression) were not to be combined. The interpretation of each HADS subscales was as follows: 0-7 normal, 8-10 mild, 11-14 moderate and 15-21 severe.
Time Frame: Baseline
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 313 | 307
units on a scale
  Anxiety total score | 3.76 (3.800) | 3.67 (3.645)
  Depression total score | 4.45 (4.081) | 4.35 (3.798)

24. Secondary Outcome: Change From Baseline in HADS Anxiety Total Score at Endpoint
Description: The HADS was a self-administered questionnaire that consisted of 2 subscales, 1 measuring anxiety (HADS-A Scale) and the other measuring depression (HADS-D Scale). Each subscale was comprised of 7 items; participants assessed how each item applied to them on a scale of 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Subscores from HADS-A (Anxiety) and HADS-D (Depression) were not to be combined. The interpretation of each HADS subscales was as follows: 0-7 normal, 8-10 mild, 11-14 moderate and 15-21 severe.
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 296 | 286
units on a scale | -0.48 (0.161) | -0.31 (0.163)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4172, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.17, 95% CI 2-sided [-0.57 to 0.24], Standard Error of Mean 0.207

25. Secondary Outcome: Change From Baseline in HADS Depression Total Score at Endpoint
Description: as for outcome 24
Time Frame: Baseline and Day 63 (Week 9)/Early Termination (Study Endpoint)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 297 | 286
units on a scale | -0.57 (0.169) | -0.38 (0.172)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.3724, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.19, 95% CI 2-sided [-0.62 to 0.23], Standard Error of Mean 0.218

ADVERSE EVENTS:
Time Frame: From Baseline till Week 10 (Day 70) and/or Early Termination.
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another, or 1 participant may have experienced both an AE and SAE during the study. All treated participants were included in the analysis.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 7/314 | 5/308
Other Adverse Events (participants affected / at risk) | 77/314 | 55/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=314) | Placebo (N=308)
Cardiac failure (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=314) | Placebo (N=308)
Vision blurred (Eye disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 5 | 0
Oedema peripheral (General disorders) | 10 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 6
Urinary tract infection (Infections and infestations) | 7 | 12
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 5
Dizziness (Nervous system disorders) | 30 | 12
Headache (Nervous system disorders) | 4 | 6
Somnolence (Nervous system disorders) | 18 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.